CLINICAL TRIAL: NCT04525092
Title: Evaluation of the Impact of Online Hemodiafiltration vs Conventional Hemodialysis in Acute Kidney Injury on Inflammatory and Clinical Outcomes
Brief Title: Online Hemodiafiltration vs Conventional Hemodialysis in Acute Kidney Injury
Acronym: HDFAKI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20.147
Record Dates: First submitted 2020-08-17; First posted 2020-08-25 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Acute Kidney Injury
Keywords: hemodialysis; hemodiafiltration; Acute kidney injury; AKI; Renal replacement therapy; Inflammation
MeSH Terms: conditions — Acute Kidney Injury; Inflammation

STUDY DESIGN:
Intervention Model Description: Pilot, Randomised, Open-label, Parallel Groups (co-intervention, 1:1:1) of three interventions: conventional HD, pre-dilution HDF and post-dilution HDF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional Hemodialysis (Active Comparator): Participants will receive intermittent HD for a minimum of 4hours per session, 3 to 4 times/week, using the 5008 High-Volume HDF Machine from Fresenius Medical Care with High Flux FX1000 Dialyzer (Mode HD).
  Interventions: Device: Conventional Hemodialysis
- Pre-dilution Hemodiafiltration (Experimental): Participants will receive intermittent pre-dilution HDF for a minimum of 4hours per session, 3 to 4 times/week, using the 5008 High-Volume HDF Machine from Fresenius Medical Care with High Flux FX1000 Dialyzer (Mode pre-dilution HDF).
  Interventions: Device: Online Pre-dilution Hemodiafiltration
- Post-dilution Hemodiafiltration (Experimental): Participants will receive intermittent post-dilution HDF for a minimum of 4hours per session, 3 to 4 times/week, using the 5008 High-Volume HDF Machine from Fresenius Medical Care with High Flux FX1000 Dialyzer (Mode post-dilution HDF).
  Interventions: Device: Online Post-dilution Hemodiafiltration

INTERVENTIONS:
Device: Online Pre-dilution Hemodiafiltration — The following parameters: maximum Blood flow rate allowed by vascular access, dialyste rate of 500 mL/min and average convective volume of >44L/session reinjected in pre-dilution mode. The dialysate composition, net ultrafiltration rate and use of anticoagulation will be prescribed according to participant's characteristics.
  Arms: Pre-dilution Hemodiafiltration
Device: Conventional Hemodialysis — Using the following parameters: maximum Blood flow rate allowed by vascular access, dialysate rate of 500 mL/min, no convection. The dialysate composition, net ultrafiltration rate and use of anticoagulation will be prescribed according to participant's characteristics.
  Arms: Conventional Hemodialysis
Device: Online Post-dilution Hemodiafiltration — The following parameters: maximum Blood flow rate allowed by vascular access, dialyste rate of 500 mL/min and average convective volume of >22L/session reinjected in pre-dilution mode. The dialysate composition and net ultrafiltration rate will be prescribed according to participant's characteristics. Usage of intra-dialysis anticoagulation is mandatory.
  Arms: Post-dilution Hemodiafiltration

SUMMARY:
Only limited data exist on the benefit of online hemodiafiltration in patient with Acute kidney injury. The objective of this pilot RCT is to assess the feasibility of a large multicentre RCT to determine whether, in patients with AKI requiring acute renal replacement therapy, does exposure to Online Hemodiafiltration reduce the inflammatory status and improve renal recovery compared to conventional intermittent hemodialysis at the ICU.

DETAILED DESCRIPTION:
Despite sparse data on the advantages of hemodiafiltration over conventional hemodialysis for intermittent dialysis, there is limited data comparing these modalities in AKI from various aetiologies in critically ill patients. As RCTs involving renal replacement therapy at the ICU are exceptionally challenging to complete, thus a rigorous RCT based on appropriate sample size and relevant clinical outcomes is crucial. The objective of this pilot RCT is to assess the feasibility of a larger multicentre RCT to determine whether, in patients with AKI requiring acute renal replacement therapy, does exposure to Post-dilution Hemodiafiltration or Pre-dilution Hemodiafiltration reduce the inflammatory status and improve renal recovery compared to conventional intermittent hemodialysis at the ICU. As post-dilution HDF has never been adequately evaluated in an ICU context, comparison between pre-dilution and post-dilution HDF is also required to confirm feasibility.

This proof-of-concept pilot trial will focus on three feasibility endpoints. It will be considered successful if the following criteria are achieved :

* Protocol adherence: If ≥85% of overall dialysis sessions are administered per-protocol according to the allocated modality
* Adherence to follow-up: If it was possible to obtain end-of-study outcomes in ≥90% of participants, and
* Participant accrual: If the average monthly enrolment is 4 or more participants per months.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised in the ICU
* Acute kidney injury stage 3 (KDIGO-AKI Criteria)
* Requiring RRT for AKI, as judged by the attending clinician (initiation) or conversion from CRRT to intermittent dialysis
* Adult of 18 years or more

Exclusion Criteria:

* Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study.
* Subjects who are participating in another study involving dialysis interventions
* Subjects or relatives/next-of-kin unable to provide written informed consent
* Creatinine clearance (CrCl) < 30 mL/min measured by 24-hour urine collection or eGFR or on chronic dialysis at baseline
* Subjects on active immunosuppressive therapy (>10mg of prednisone, biologic therapies, calcineurin inhibitors, mTOR inhibitors or antimetabolites)
* Subjects with active contraindication to anticoagulation during dialysis session
* Subjects whose RRT is not part of their life goal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Protocol adherence (feasibility) | 90 days
  If ≥85% of overall dialysis sessions are administered per-protocol according to the allocated modality
Adherence to follow-up (feasibility) | 90 days
  If it was possible to obtain end-of-study outcomes in ≥90% of participants
Participant accrual (feasibility) | 90 days
  If the average monthly enrolment is 4 or more participants per months

SECONDARY OUTCOMES:
Mortality | 30 days
  (overall mortality)
Mortality | 90 days
  (overall mortality)
End-of-study eGFR | 90 days
  (mL/min/1.73m2)
Dialysis dependence | 90 days
  Defined as the receipt of dialysis at day 90
Total number of days on dialysis | 90 days
  (in patients with renal recovery)
Length of hospitalisation stay | 90 days
  (days)
Number of patients with hemodynamic instability during dialysis treatment (first week) | 7 days
  (using two definitions):
  * Defined as systolic blood pressure drop <90 mmHg requiring intervention (one of the following: increase of vasopressor, Ultrafiltration cessation/reduction, termination of the dialysis session or fluid bolus)
  * Variations in the vasoactive-inotropic score between pre-dialysis and per-dialysis timepoint
Number of dialysis session complicated by Circuit/filter clotting | 90 days
  (proportion)

OTHER OUTCOMES:
(Exploratory) Inflammatory serum biomarkers modulation | Day 0 and Day 7
  (Percentage of reduction by clearance of the following biomarkers: C-reactive protein, CCL11, CCL26, Fibroblast growth Factor, GM-CSF, ICAM-1, IFN-γ, IL-10, IL-12/IL-23p40, IL-12p70, IL-13, IL-15, IL-16, IL-17A, IL-1α, IL-1β, IL 2, IL-4, IL-5, IL-6, IL-7, CXCL8, CXCL10, CCL2, CCL3, CCL4, CCL13, CCL22, Placental growth factor, Serum Amyloid A, CCL17, Tyrosine kinase 2 (Tie)-2, TNF-α, TNF-β, VCAM-1 and VEGF)
(Exploratory) Phenotype of circulation neutrophils | Day 0 and Day 7
  Activation phenotype of circulating neutrophils, using variation in the mean fluorescent intensity (MFI) by flux-cytometry, measured at randomisation (Day0) and after first week of treatment (Day7)
(Exploratory) Phenotype of circulation monocytes | Day 0 and Day 7
  Activation phenotype of circulating monocytes, using variation in the mean fluorescent intensity (MFI) by flux-cytometry, measured at randomisation (Day0) and after first week of treatment (Day7)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Maxime Cote, MD, MSc, Principal Investigator — CHUM
Locations (2):
- Centre de recherche du CHUM, Montreal, Quebec, Canada
- Clinical Research Centre University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No